CLINICAL TRIAL: NCT02557958
Title: Chronic Obstructive Pulmonary Disease Transcription Factor and Cytokine Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-0769
Record Dates: First submitted 2015-09-02; First posted 2015-09-23 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Azithromycin (Experimental): Azithromycin 250mg daily, single daily use for 8 weeks
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): Placebo daily for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — We hypothesize that in patients with COPD, treatment with azithromycin will show reduced inflammatory markers, transcription factors changes, and lung function changes consistent with reduced inflammation.
  Other Names: Zithromax
  Arms: Azithromycin
Drug: Placebo — We hypothesize that in patients with COPD, treatment with placebo will show NO change in inflammatory markers, transcription factor changes and lung function from baseline.
  Arms: Placebo

SUMMARY:
Chronic Obstructive Pulmonary Disease Transcription Factor and Cytokine Study.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is the 4th leading cause of death in the United States. It is projected to be the leading cause of death by 2020. As many as 24 million Americans are estimated to suffer from impaired lung function. Of those more than 12 million were actually diagnosed with COPD, and over 118,000 deaths were attributed to COPD in 2004.

COPD has been linked with an increased risk for lung cancer. Both airway obstruction, defined by abnormal pulmonary function tests (PFTs), and CT scan diagnosed emphysema were shown to be independent risk factors for lung cancer.

Treatment for COPD includes cessation of environmental exposures (i.e. smoking), dampening the inflammatory response, symptoms control and, for a small subgroup, surgical approaches and lung transplant. Nevertheless, the effectiveness of these treatment options to change the natural history of this disease is very limited. Recent evidence suggests a new role for macrolides as immune-modulators in patients with COPD, although the mechanisms are not clearly determined.

The investigators hypothesize that in patients with COPD, treatment with azithromycin will show reduced inflammatory markers, transcription factors changes, and lung function changes consistent with reduced inflammation.

ELIGIBILITY:
* Key Inclusion Criteria: List primary criteria for study inclusion (i.e. do not need to enter entire list of inclusion criteria).

  1. Patient must be 50 years old or older.
  2. Patient must have a smoking history of at least 20 pack-years
  3. Patient must have stable COPD, GOLD 0, I and/or IIA.
  4. CT of chest with evidence of emphysema
* Key Exclusion Criteria: List primary criteria for study exclusion (i.e. do not need to enter entire list of inclusion criteria).

  1. FEV1 < 70%.
  2. Exacerbations (defined as use of oral steroids or antibiotics) in the previous month.
  3. Cardiovascular Disease defined as abnormal EKG, known or suspected coronary artery disease or congestive heart failure.
  4. Diabetes mellitus
  5. Renal disease
  6. Liver disease
  7. Lung cancer
  8. ETOH use of more than >6 beers >4 mixed drinks daily

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Inflammatory markers | outcome will be assessed up to two months post initial bronchoscopy
  Cytokines in BAL in pg/mL

SECONDARY OUTCOMES:
transcription factor changes | outcome will be assessed up to two months post initial bronchoscopy
  BAL cell differential in percentage
Lung function changes | outcome will be assessed up to two months post initial bronchoscopy
  Forced Vital Capacity (FVC)

REFERENCES:
- [Derived] Segal LN, Clemente JC, Wu BG, Wikoff WR, Gao Z, Li Y, Ko JP, Rom WN, Blaser MJ, Weiden MD. Randomised, double-blind, placebo-controlled trial with azithromycin selects for anti-inflammatory microbial metabolites in the emphysematous lung. Thorax. 2017 Jan;72(1):13-22. doi: 10.1136/thoraxjnl-2016-208599. Epub 2016 Aug 2. PMID 27486204